CLINICAL TRIAL: NCT00854308
Title: A Randomized, Phase II, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Activity of MetMAb, a Monovalent Antagonist Antibody to the Receptor Met, Administered to Patients With Advanced Non-Small Cell Lung Cancer, in Combination With Tarceva (Erlotinib)
Brief Title: A Study of MetMAb Administered to Patients With Advanced Non-Small Cell Lung Cancer, in Combination With Tarceva (Erlotinib)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAM4558g
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2011-10-18 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2012-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tarceva; Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; onartuzumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MetMAb + Erlotinib (Experimental): MetMab 15 mg/kg intravenous (IV) infusion every 3 weeks + Erlotinib 150 mg orally once daily until progression of disease or unacceptable toxicity.
  Interventions: Drug: Erlotinib HCl; Drug: MetMAb
- Placebo + Erlotinib (Placebo Comparator): Placebo IV infusion every 3 weeks + Erlotinib 150 mg orally daily until progression of disease or unacceptable toxicity.
  Interventions: Drug: Erlotinib HCl; Drug: placebo (0.9 % saline)

INTERVENTIONS:
Drug: Erlotinib HCl — Erlotinib 150 mg oral dose once daily.
  Other Names: Tarceva
Drug: MetMAb — MetMab (a monovalent antagonist antibody to the receptor MET) 15 mg/kg in 250 CC 0.9% saline intravenous infusion every 3 weeks.
  Arms: MetMAb + Erlotinib
Drug: placebo (0.9 % saline) — Placebo Intravenous infusion every 3 weeks.
  Arms: Placebo + Erlotinib

SUMMARY:
This is a Phase II, double-blind, randomized, multicenter trial designed to preliminarily evaluate the activity and safety of treatment with MetMAb + erlotinib versus erlotinib + placebo in second- and third-line Non-Small Cell Lung Cancer (NSCLC). Up to 180 patients will be randomized in a 1:1 ratio to one of the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Histologically confirmed NSCLC
* Availability of a tumor specimen
* Recurrent or progressive disease following at least one chemo containing regimen for Stage IIIB/IV disease
* Measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST)
* At least one measurable lesion on a pre-treatment 18-fluorodeoxyglcose-positron emission tomography (FDG-PET) scan that is also a target lesion on computed tomography (CT) according to RECIST

Exclusion Criteria:

* More than two prior treatments for Stage IIIB/IV
* More than 30 days of exposure to an investigational or marketed agent that can act by EGFR inhibition, or a known epidermal growth factor receptor (EGFR)-related toxicity resulting in dose modifications
* Chemotherapy, biologic therapy, radiotherapy or investigational drug within 28 days prior to randomization
* Untreated and/or active (progressing or requiring anticonvulsants or corticosteroids for symptomatic control) central nervous system (CNS) metastasis
* History of serious systemic disease within the past 6 months prior to randomization
* Uncontrolled diabetes
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization
* Anticipation of need for a major surgical procedure during the course of the study
* Local palliative radiotherapy within 7 days prior to randomization or persistent adverse effects from radiotherapy that have not been resolved to Grade II or less prior to randomization
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premal Patel, M.D., Ph.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-seven patients in the placebo + erlotinib arm with disease progression in the blinded treatment stage elected to receive MetMAb + erlotinib in the optional open-label phase of the study.
Groups:
- MetMAb + Erlotinib: MetMab (a monovalent antagonist antibody to the receptor MET) 15 mg/kg intravenous (IV) infusion every 3 weeks + Erlotinib 150 mg orally once daily until progression of disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Started | 69 | 68
Received Study Drug | 69 | 67
Completed | 7 (Completed participants in both arms were still receiving study drug when analyses were performed.) | 1
Not Completed | 62 | 67
Not completed — Disease progression | 42 | 50
Not completed — Adverse Event | 8 | 3
Not completed — Death | 2 | 5
Not completed — Physician Decision | 6 | 6
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Sponsor's decision to terminate study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.4) | 62.7 (10.6) | 63.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the first occurrence of progression or relapse (as per Response Evaluation Criteria in Solid Tumors (RECIST 1.0) and assessed by the site radiologist or investigator) or death on study from any cause (within 30 days of last treatment).
Time Frame: Time from randomization to the first occurrence of progression/relapse or death on study. (Up to 20 months)
Population: All randomized intent-to-treat patients.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Number analyzed (Participants) | 69 | 68
months | 2.2 [1.38 to 2.86] | 2.6 [1.45 to 2.76]
Statistical Analysis 1: Comparison: MetMAb + Erlotinib vs Placebo + Erlotinib; The null hypothesis is that there is no difference in PFS between MetMab + Erlotinib and Placebo + Erlotinib. The alternate hypothesis is that MetMab + Erlotinib would have prolonged PFS compared with Placebo + Erlotinib; Test type: Superiority or Other; p = 0.6873, Log Rank; Hazard Ratio (HR) = 1.086, 95% CI 2-sided [0.727 to 1.622] — The hazard ratio was estimated using Cox Regression and was stratified for smoking status, Eastern Cooperative Oncology Group (ECOG) performance status and histology. The hazard ratio is relative to Placebo + Erlotinib

2. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response (partial and complete response as determined using RECIST 1.0).
  Partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter.
  Complete response was defined as disappearance of all target lesions.
Time Frame: Start of treatment until disease progression/recurrence or death on study. (Up to 20 months)
Population: All randomized intent-to-treat patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Number analyzed (Participants) | 69 | 68
Percentage of participants | 5.8 [2.0 to 13.9] | 4.4 [1.2 to 11.7]
Statistical Analysis 1: Comparison: MetMAb + Erlotinib vs Placebo + Erlotinib; The null hypothesis is that there is no difference in Objective Response between MetMab + Erlotinib and Placebo + Erlotinib. The alternate hypothesis is that MetMab + Erlotinib would have better Objective Response compared with Placebo + Erlotinib; Test type: Superiority or Other; p = 0.7101, Cochran-Mantel-Haenszel — P-value was stratified for smoking status, ECOG performance status and histology

3. Secondary Outcome: Percentage of Participants With Objective Response in Patients With Met Diagnostic-Positive Tumors
Description: Objective response (OR); partial and complete response as determined using RECIST 1.0 in patients with Met Diagnostic-Positive Tumors as determined by immunohistochemistry.
  Partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter.
  Complete response was defined as disappearance of all target lesions.
Time Frame: Start of treatment until disease progression/recurrence or death on study. (Up to 20 months)
Population: All randomized intent-to-treat patients with Met Diagnostic-positive tumors.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Number analyzed (Participants) | 35 | 31
Percentage of participants | 8.6 [2.4 to 21.5] | 3.2 [0.2 to 16.1]
Statistical Analysis 1: Comparison: MetMAb + Erlotinib vs Placebo + Erlotinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3671, Cochran-Mantel-Haenszel — P-value was stratified for smoking status, ECOG performance status and histology

4. Primary Outcome: Progression-free Survival in Patients With Met Diagnostic-Positive Tumors
Description: Progression-free survival (PFS) in participants with Met Diagnostic-Positive tumors as determined by immunohistochemistry.
  PFS was defined as the time from randomization to the first occurrence of progression or relapse (as per Response Evaluation Criteria in Solid Tumors (RECIST 1.0) and assessed by the site radiologist or investigator) or death on study from any cause (within 30 days of last treatment).
Time Frame: Time from randomization to the first occurrence of progression/relapse or death on study. (Up to 20 months)
Population: All randomized intent-to-treat patients with Met Diagnostic-Positive tumors.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Number analyzed (Participants) | 35 | 31
months | 2.9 [1.38 to 6.21] | 1.5 [1.35 to 2.63]
Statistical Analysis 1: Comparison: MetMAb + Erlotinib vs Placebo + Erlotinib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0418, Log Rank; Hazard Ratio (HR) = 0.529, 95% CI 2-sided [0.284 to 0.986] — The hazard ratio was estimated using Cox Regression and was stratified for smoking status, ECOG performance status and histology. The hazard ratio is relative to Placebo + Erlotinib

5. Secondary Outcome: Duration of Overall Response
Time Frame: Date of initial response until date of progression or death on study. (Up to 20 months)
Population: All randomized intent-to-treat patients. Analyses of duration of response were not performed because of the small number of patients with objective responses.
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 20 months
Arm/Group | MetMAb + Erlotinib | Placebo + Erlotinib
Serious Adverse Events (participants affected / at risk) | 29/69 | 22/67
Other Adverse Events (participants affected / at risk) | 68/69 | 67/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MetMAb + Erlotinib (N=69) | Placebo + Erlotinib (N=67)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 1 | 0
DEATH (General disorders) | 0 | 1
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0
PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 4 | 1
LUNG INFECTION (Infections and infestations) | 1 | 1
CELLULITIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
DELIRIUM (Psychiatric disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
EMBOLISM VENOUS (Vascular disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MetMAb + Erlotinib (N=69) | Placebo + Erlotinib (N=67)
ANAEMIA (Blood and lymphatic system disorders) | 10 | 10
DIARRHOEA (Gastrointestinal disorders) | 28 | 35
NAUSEA (Gastrointestinal disorders) | 22 | 21
VOMITING (Gastrointestinal disorders) | 4 | 13
DYSPEPSIA (Gastrointestinal disorders) | 5 | 6
CONSTIPATION (Gastrointestinal disorders) | 4 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 2
STOMATITIS (Gastrointestinal disorders) | 4 | 3
FATIGUE (General disorders) | 22 | 24
OEDEMA PERIPHERAL (General disorders) | 16 | 5
PYREXIA (General disorders) | 10 | 6
ASTHENIA (General disorders) | 9 | 6
PAIN (General disorders) | 4 | 8
CHEST PAIN (General disorders) | 2 | 7
OEDEMA (General disorders) | 6 | 2
URINARY TRACT INFECTION (Infections and infestations) | 4 | 6
PNEUMONIA (Infections and infestations) | 5 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 14 | 16
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 4
DIZZINESS (Nervous system disorders) | 5 | 6
DYSGEUSIA (Nervous system disorders) | 3 | 4
HEADACHE (Nervous system disorders) | 2 | 4
ANXIETY (Psychiatric disorders) | 6 | 7
INSOMNIA (Psychiatric disorders) | 8 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 16
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 | 13
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 6 | 5
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 1
RASH (Skin and subcutaneous tissue disorders) | 42 | 41
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 10 | 10
DRY SKIN (Skin and subcutaneous tissue disorders) | 8 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 8
HYPOTENSION (Vascular disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.